CLINICAL TRIAL: NCT05328635
Title: The Effect of Multidisciplinary Intervention on Patients With Persistent Post-traumatic Headache
Brief Title: Post-traumatic Headache Multidisciplinary Study
Acronym: PTHMS
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Principal investigator, MD and associate professor, Danish Headache Center
Other Study IDs: DanishHC180322
Record Dates: First submitted 2022-03-18; First posted 2022-04-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Post-Traumatic Headache; Post-Concussion Syndrome
MeSH Terms: conditions — Post-Traumatic Headache; Post-Concussion Syndrome | interventions — candesartan; Amitriptyline; Gabapentin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Candesartan — Multdisciplinary approach
  Other Names: Amitriptylin; Gabapentin

SUMMARY:
The study will investigate the effect of pharmacological preventive treatment, education, physiotherapy and psychological counselling on the headache and associated symptoms in patients refered to the Danish Headache Center

DETAILED DESCRIPTION:
Pharmacological interventions are candesartan, amitritylin and gabapentin depending on the headache phenotype. In total 3 visits spanned over 1 year

Education is conducted as group sessions of up to 10 patients by two specialist nurses 2 x 90 min Physiotherapy is conducted as group sessions of up to 5 patients by physiotherapists 8 x 60 min plus 2 individual sessions.

Psychology is conducted as group sessions of up to 10 patients by psychologist 3x60 min plus option of 1 individual session.

ELIGIBILITY:
Inclusion Criteria:

Patients with post-traumatic headache

-

Exclusion Criteria:

* Medication-overuse headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a head trauma as a cause of the headache will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in headache days | 1 year
  Headache days will be obtained via a validated questionaire
Rivermead post-concussion questionare score | 1 year
  Rivermead is a validated questionaire to assess concussion symptoms
HADS-scores | 1 year
  HADS = Hospital anxiety and depression scale. A validated tool to assesss depression and anxiety symptoms
Self-perceived health | 1 year
  based on EU-SILC validated question on self-perceived health ('How is your health in general?'), which contains five answering categories; 1) very good, 2) good, 3) fair, 4) bad, 5) very bad.
Level of physical activity | 1 year
  Based on questionaire, where patients can choose: Low level of physical activity: primarily sedentary activities or light exercise at least 4 hours a week, or

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No